CLINICAL TRIAL: NCT03704116
Title: Project Expedition: Executive Function Training Intervention for Chronic Traumatic Brain Injury
Brief Title: Executive Function Training Intervention for Chronic Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Applied Research Associates, Inc (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Krawczyk, Professor, Debbie and Jim Francis Chair, The University of Texas at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTDallas
Record Dates: First submitted 2018-07-03; First posted 2018-10-12 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Traumatic Brain Injury
Keywords: chronic traumatic brain injury; cognition; executive function
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — CHE protein, Arabidopsis

STUDY DESIGN:
Intervention Model Description: Two groups run in parallel (active and control)
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expedition: Strategic Advantage (Active Comparator): Software-based intervention simulating daily life cognitive challenges. Delivered 1 hour per day, 5 days per week for 4 weeks. Includes 8 check-in phone calls with an experimenter. Includes escalating challenge levels.
  Interventions: Behavioral: Expedition
- Expedition: Informational Advantage (Placebo Comparator): Software-based intervention simulating daily life cognitive challenges. Delivered 1 hour per day, 5 days per week for 4 weeks. Includes 8 check-in phone calls with an experimenter. Includes capped challenge levels.
  Interventions: Behavioral: Expedition

INTERVENTIONS:
Behavioral: Expedition — On a laptop computer participants work on simulated daily life activities including packing for a trip, navigating a transit system, and learning at museum attractions. The intervention increases difficulty as participants accomplish goals. We are testing the effects of this performance challenge on executive function measures.

SUMMARY:
Traumatic Brain Injury (TBI) is a prevalent disorder developed by military personnel. While some individuals recover function within months after injury, others continue to suffer from cognitive problems months to years later and may not become evident immediately, particularly for the recently transitioned veteran. Chronic TBI cases may include persistent difficulties in cognition that negatively impact employment and personal relationships.

The investigators will test and evaluate software-based interventions aimed at improving cognition in veterans experiencing everyday life cognitive deficits due to TBI. The interventions will be administered on a computer using a tele-health approach. Two conditions will be compared, an active condition challenging memory, inhibitory control and planning, and a context-matched control condition that is lower on these challenge levels.

DETAILED DESCRIPTION:
The investigators will evaluate the improvement of chronic TBI symptoms after interventions. The investigators will evaluate the improvement of chronic mTBI symptoms using Magnetic Resonance Imaging (MRI)-based injury markers, cognitive functions, and real-world functioning questionnaires.

The investigators will recruit military veterans with mild-to-moderate chronic TBI (at least 3 months post injury). The investigators will gather neuropsychological, cognitive, and neuroimaging (functional MRI, resting-state functional MRI) measures. The efficacy of the active compared to control intervention will be evaluated in 100 chronic TBI veterans. All participants will be randomized to a group to complete four weeks of intervention over 20 performance sessions. Over the course of training participants will face escalating challenges in each of these domains, thereby improving their overall skills. The software captures response times and accuracy of performance throughout each task. Evaluations of cognition (neuropsychological testing), brain (MRI), real life functional ability (survey data), and real life performance data (multiple errands tasks) will be gathered pre- and post-intervention to evaluate cognitive, brain-based, and real life functional improvements.

ELIGIBILITY:
Inclusion Criteria:

* male and female military veteran adults between the ages of 19 to 55 years (served in the military (any branch))
* who have sustained a traumatic brain injury at least 3 months previously
* who can comprehend simple instructions, perform the tests, and take part in the intervention training
* Selection criteria will also include participants who can safely have an MRI, who can tolerate at least 2 hours of intervention sessions at a time, and who can participate in tasks involving motor abilities such as use of at least one arm and hand
* No racial/ethnic groups will be excluded, although the patients must be able to speak, read, and comprehend English well enough to participate in the testing and treatment sessions, since the assessments are not normed or translated in other languages at this time.
* Also, we will screen for possible Post Traumatic Stress Disorder (PTSD) using the Mississippi PTSD Questionnaire, but it will not be an exclusionary criteria.

Exclusion Criteria:

* someone who is not proficient in reading, comprehending, and speaking English,
* has pre-existing cerebral palsy, mental retardation, autism, epilepsy, schizophrenia, or pervasive developmental disorder.
* Individuals with psychosis, active behavioral disorder, or uncontrolled epilepsy will be excluded.
* Pregnant women will be excluded, since the effects of the treatment or the procedures on a fetus are unknown.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Virtual Multiple Errands Test | change is evaluated from the beginning of the intervention to after completion (1 month in between)
  executive function measure carried out in computer simulation of shopping market

SECONDARY OUTCOMES:
Resting-State functional Magnetic Resonance Imaging (fMRI) | change is evaluated from the beginning of the intervention to after completion (1 month in between)
  functional connectivity assessment
Task-based functional Magnetic Resonance Imaging (fMRI) | change is evaluated from the beginning of the intervention to after completion (1 month in between)
  functional brain imaging attention task
Automated Neuropsychological Assessement Metrics (ANAM) | change is evaluated from the beginning of the intervention to after completion (1 month in between)
  code substitution, go/no go, logical relations, manikin, match-to-sample, Mathematical processing
Traumatic Brain Injury (TBI) Awareness Questionnaire | change is evaluated from the beginning of the intervention to after completion (1 month in between)
  Survey measure asking for estimate of current symptoms compared to before brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Clover, Study Director — Applied Research Associates
Locations (1):
- The University of Texas at Dallas Center for BrainHealth, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krawczyk DC, Han K, Martinez D, Rakic J, Kmiecik MJ, Chang Z, Nguyen L, Lundie M, Cole RC, Nagele M, Didehbani N. Executive function training in chronic traumatic brain injury patients: study protocol. Trials. 2019 Jul 15;20(1):435. doi: 10.1186/s13063-019-3526-x. PMID 31307502

DOCUMENTS (2):
  • Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03704116/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT03704116/SAP_001.pdf